CLINICAL TRIAL: NCT04585919
Title: Paired Promotion of Colorectal Cancer and Social Determinants of Health Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Karen Emmons, Professor of Social and Behavioral Sciences, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: 67702115; P50CA244433 (NIH)
Record Dates: First submitted 2020-09-30; First posted 2020-10-14 (Actual); Results first posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Colorectal Cancer; Social Determinants of Health
Keywords: implementation science; colorectal cancer screening; social determinants of health screening
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: This trial uses a randomized stepped wedge study design. This pragmatic design involves a sequential, randomized roll-out of the intervention across the four participating clinical sites or "clusters" over 8 week intervals or "steps." The intervention is the paired outreach to patients in need of CRC screening to offer FIT screening and screening for SDOH. The participants who will be enrolled are CHC staff who will provide input on the implementation processes and outcomes.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paired Screening Intervention (Experimental)
  Interventions: Behavioral: Paired Screening Intervention
- Usual Care Control (No Intervention): In this stepped wedge design, all sites have a period of being in usual care, and then providing the Paired Screening Intervention. Sites serve as their own controls in this design.

INTERVENTIONS:
Behavioral: Paired Screening Intervention — The intervention is the implementation of a paired outreach strategy to patients in need of colorectal cancer screening to offer FIT testing and to complete screening for social determinants of health. These screening activities are part of routine practice but the intervention that is being implemented is the paired outreach for both CRC screening and SDOH screening.
  Arms: Paired Screening Intervention

SUMMARY:
This work is an implementation science study that examines different aspects of implementing a single intervention. The intervention consists of asking community health centers to implement an outreach strategy to screen patients for colorectal cancer and for social determinants of health in community health centers at the same contact point. These are both clinical targets that the CHCs feel that their patients need and want to offer at a higher rate. The intervention consists of outreach to patients in need of colorectal cancer screening (CRC) to offer fecal immunochemical test (FIT) screening and screening for social determinants of health (SDOH). In this implementation science study, the intervention is an evidence-based intervention being implemented in real-world clinical practice. The intervention is the outreach to offer FIT and SDOH, conducted by clinic staff. Both evidence-based screening activities-FIT and SDOH screening-are used in the practices included in the study but pairing them is intended to increase efficiency and patient-centeredness by addressing health related social needs that may impact patients' ability to engage in cancer screening. The study aims to test the effect of implementing the intervention on clinical and process outcomes. Clinical outcomes are CRC screening and SDOH screening. Analysis of process outcomes includes measuring what organizational factors influence implementation.

ELIGIBILITY:
Study participants include community health center staff participating in interviews about the implementation of the intervention. Up to four community health center staff members at each of the four community health centers will participate in key informant interviews twice per year. Patients will receive the paired screening intervention as part of their routine care and will not be individually recruited for the study because the intervention is being offered as part of routine care.

Staff Participants

Inclusion Criteria:

* Staff from community health centers who facilitate screening
* Age 18 and older

Exclusion Criteria:

* Have not participated in the implementation of the paired screening intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Emmons, PhD, Principal Investigator — Harvard TH Chan School of Public Health
Locations (4):
- United States (4):
  - Harbor Health Services, Boston, Massachusetts
  - Brockton Neighborhood Health Center, Brockton, Massachusetts
  - Lowell Community Health Center, Lowell, Massachusetts
  - Manet Community Health Center, Quincy, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported here, after deidentification (text, tables, figures, and appendices). Upon request and appropriate approvals.
Time Frame: 6 months after publication, and for 3 years.
Access Criteria: Outside investigators will need an approved concept proposal to analyze study data and spend the requisite time with study staff to learn about the data elements needed to conduct the proposed analysis. With the assistance of our analytic team, s/he will draft a detailed analysis plan and present to the core group of co-investigators. The discussion at this meeting ensures adequate knowledge of the data, and the presenter gains much insight into how the analysis can be most useful and how it relates to previous analyses. Once the plan is approved by this group, it must also be approved by the CHCs that provide the de-identified data. Following approval by the appropriate IRBs and confirmation that it meets HIPAA requirements, s/he may sign a DUA to use a secure, de-identified dataset to complete only the approved analyses and write the manuscript(s) offsite. A formal data analysis plan application and DUA are still in development. Requests should be directed to jdaly@hsph.harvard.edu.

REFERENCES:
- [Derived] Kruse GR, Percac-Lima S, Barber-Dubois M, Davies ME, Gundersen DA, Ho O, Mascioli L, Munshi M, Perry S, Singh D, Thomas A, Emmons KM, Haas JS. Bundling Colorectal Cancer Screening Outreach with Screening for Social Risk in Federally Qualified Health Centers: A Stepped-Wedge Implementation-Effectiveness Study. J Gen Intern Med. 2024 May;39(7):1188-1195. doi: 10.1007/s11606-024-08654-5. Epub 2024 Feb 8. PMID 38332440
- [Derived] Aschbrenner KA, Kruse G, Emmons KM, Singh D, Barber-Dubois ME, Miller AM, Thomas AN, Bartels SJ. Stakeholder and Equity Data-Driven Implementation: a Mixed Methods Pilot Feasibility Study. Prev Sci. 2024 Apr;25(Suppl 1):136-146. doi: 10.1007/s11121-022-01442-9. Epub 2022 Oct 4. PMID 36194312

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants include community health center staff participating in interviews about the implementation of the intervention. Patients received the paired screening intervention as part of their routine care and were not individually recruited for the study because the intervention was offered as part of routine care.
Pre-assignment Details: Community health center staff are only considered enrolled.
Units Other Than Participants: Community Health Center
Groups:
- Sequence A: 8 months usual care, then 4 months paired outreach followed by 10 months planned adaptation.
  Paired Screening Intervention: The intervention is the implementation of a paired outreach strategy to patients in need of colorectal cancer screening to offer FIT testing and to complete screening for social determinants of health. These screening activities are part of routine practice but the intervention that is being implemented is the paired outreach for both CRC screening and SDOH screening.
  In this stepped wedge design, all sites have a period of being in usual care, and then providing the Paired Screening Intervention. Sites serve as their own controls in this design.
- Sequence B: 10 months Usual care, then 4 months paired outreach, followed by 8 months planned adaptation.
  Paired Screening Intervention: The intervention is the implementation of a paired outreach strategy to patients in need of colorectal cancer screening to offer FIT testing and to complete screening for social determinants of health. These screening activities are part of routine practice but the intervention that is being implemented is the paired outreach for both CRC screening and SDOH screening.
  In this stepped wedge design, all sites have a period of being in usual care, and then providing the Paired Screening Intervention. Sites serve as their own controls in this design.
- Sequence C: 12 months usual care, then 4 months paired outreach followed by 6 months planned adaptation.
  Paired Screening Intervention: The intervention is the implementation of a paired outreach strategy to patients in need of colorectal cancer screening to offer FIT testing and to complete screening for social determinants of health. These screening activities are part of routine practice but the intervention that is being implemented is the paired outreach for both CRC screening and SDOH screening.
  In this stepped wedge design, all sites have a period of being in usual care, and then providing the Paired Screening Intervention. Sites serve as their own controls in this design.
- Sequence D: 14 months Usual care, then 4 months paired outreach followed by 4 months planned adaptation.
  Paired Screening Intervention: The intervention is the implementation of a paired outreach strategy to patients in need of colorectal cancer screening to offer FIT testing and to complete screening for social determinants of health. These screening activities are part of routine practice but the intervention that is being implemented is the paired outreach for both CRC screening and SDOH screening.
  In this stepped wedge design, all sites have a period of being in usual care, and then providing the Paired Screening Intervention. Sites serve as their own controls in this design.
Period: Usual Care
Arm/Group | Sequence A | Sequence B | Sequence C | Sequence D
Started (Number of community health center staff) | 7; 1 Community Health Center | 6; 1 Community Health Center | 9; 1 Community Health Center | 4; 1 Community Health Center
Number of Patients (Patients are not enrolled) | 5947; 1 Community Health Center | 7652; 1 Community Health Center | 7311; 1 Community Health Center | 6317; 1 Community Health Center
Completed | 7; 1 Community Health Center | 6; 1 Community Health Center | 9; 1 Community Health Center | 4; 1 Community Health Center
Not Completed | 0; 0 Community Health Center | 0; 0 Community Health Center | 0; 0 Community Health Center | 0; 0 Community Health Center
Period: Paired Outreach
Arm/Group | Sequence A | Sequence B | Sequence C | Sequence D
Started (Number of community health center staff) | 7; 1 Community Health Center | 6; 1 Community Health Center | 9; 1 Community Health Center | 4; 1 Community Health Center
Number of Patients (Patients are not enrolled) | 6453; 1 Community Health Center | 13401; 1 Community Health Center | 7272; 1 Community Health Center | 6254; 1 Community Health Center
Completed | 7; 1 Community Health Center | 6; 1 Community Health Center | 9; 1 Community Health Center | 4; 1 Community Health Center
Not Completed | 0; 0 Community Health Center | 0; 0 Community Health Center | 0; 0 Community Health Center | 0; 0 Community Health Center

BASELINE CHARACTERISTICS:
Population: Demographic data were not collected from participants (i.e., community health center staff) described in Participant Flow. Patients received the paired screening intervention as part of their routine care and were not individually recruited for the study because the intervention is being offered as part of routine care. Baseline characteristics and outcomes reported are based on the patient-level data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Paired Screening Intervention | Usual Care Control | Total
Number analyzed (Participants) | 33380 | 27227 | 60607
Age, Continuous [Mean (Standard Deviation); unit: years] — unique patient count in each arm
  years | 61.4 (6.9) | 61.6 (6.8) | 61.5 (6.9)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 17906 | 14381 | 32287
  Male | 15460 | 12845 | 28305
  Other | 14 | 1 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3644 | 3188 | 6832
  Not Hispanic or Latino | 25184 | 20536 | 45720
  Unknown or Not Reported | 4552 | 3503 | 8055
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 83 | 63 | 146
  Asian | 3381 | 2844 | 6225
  Native Hawaiian or Other Pacific Islander | 166 | 139 | 305
  Black or African American | 6843 | 6311 | 13154
  White | 17612 | 13414 | 31026
  More than one race | 562 | 496 | 1058
  Unknown or Not Reported | 4733 | 3960 | 8693

OUTCOME MEASURES:

1. Primary Outcome: Conditional Odds Ratio of Patients Screened for Colorectal Cancer During Intervention Compared to Patients Screened During Usual Care
Description: Colorectal cancer screening completion by any guideline-based method. Adjusting for patient socio-demographics, comorbidities, number of healthcare visits, and secular trend. Documented screening in EHR for patients unscreened at the beginning of the step.
Time Frame: 13 pre implementation months, 14 post-implementation months
Population: 4 Community health centers were randomized to a sequence of implementation start and each observed for an average of 2.5 control periods (stepped wedge steps) and 5.5 intervention periods (stepped wedge steps).
Measure: Number; unit: Conditional odds
Units Other Than Participants: health centers
Arm/Group | Paired Screening Intervention | Usual Care Control
Number analyzed (Participants) | 33380 | 27227
Number analyzed (health centers) | 4 | 4
Conditional odds | 0.068 | 0.028
Statistical Analysis 1: Comparison: Paired Screening Intervention vs Usual Care Control; Test type: Superiority; p = 0.005, Mixed Models Analysis; Generalized linear mixed effect model controlling for secular trend, patient sociodemographic and health characteristics

2. Primary Outcome: Conditional Odds Ratio of Patients Screened for Social Needs During Intervention Compared to Patients Screened During Usual Care
Description: Completion of social needs screening (collected as part of routine clinical care). Adjusting for patient socio-demographics, comorbidities, number of healthcare visits, and secular trend. Documented screening in EHR for patients unscreened at the beginning of the step.
Time Frame: 13 pre implementation months, 14 post-implementation months
Population: as for outcome 1
Measure: Number; unit: Conditional odds
Units Other Than Participants: health centers
Arm/Group | Paired Screening Intervention | Usual Care Control
Number analyzed (Participants) | 33380 | 27227
Number analyzed (health centers) | 4 | 4
Conditional odds | 0.213 | 0.333
Statistical Analysis 1: Comparison: Paired Screening Intervention vs Usual Care Control; Test type: Superiority; p = 0.19, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Number of FIT Kits Mailed
Description: Adoption measured by number of FIT kits mailed to patients. Data were summed to calculate a single value.
Time Frame: 4 months post-implementation, 8 months post-implementation
Measure: Number; unit: FIT kits
Units Other Than Participants: health centers
Arm/Group | Paired Screening Intervention
Number analyzed (Participants) | 25599
Number analyzed (health centers) | 4
FIT kits | 4404

4. Secondary Outcome: Number of Reminders Per FIT Mailing
Description: Adoption measured by number of reminders per FIT mailing to patients. Data were summed to calculate a single value.
Time Frame: 4 months post-implementation, 8 months post-implementation
Population: unique patients within the 4 months post-implementation, 8 months post-implementation
Measure: Number; unit: reminders per mailed FIT kits
Units Other Than Participants: health centers
Arm/Group | Paired Screening Intervention
Number analyzed (Participants) | 25599
Number analyzed (health centers) | 4
reminders per mailed FIT kits | 0.87

5. Secondary Outcome: Number of Reminders Per FIT Return
Description: Adoption measured by number of reminders per FIT returned. Data were summed to calculate a single value.
Time Frame: 4 months post-implementation, 8 months post-implementation
Measure: Number; unit: reminders per returned FIT kit
Units Other Than Participants: health centers
Arm/Group | Paired Screening Intervention
Number analyzed (Participants) | 25599
Number analyzed (health centers) | 4
reminders per returned FIT kit | 11.7

ADVERSE EVENTS:
Description: Patients received the paired screening intervention as part of their routine care and were not individually recruited for the study because the intervention was offered as part of routine care. Enrolled study participants were community health center staff participating in interviews about the implementation of the intervention. Therefore adverse event reporting did not apply.
Arm/Group | Paired Screening Intervention | Usual Care Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-09): https://cdn.clinicaltrials.gov/large-docs/19/NCT04585919/Prot_SAP_000.pdf